CLINICAL TRIAL: NCT05658133
Title: Understanding Sports Nutrition Knowledge of High School Athletes and Influencers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-2109
Record Dates: First submitted 2022-12-09; First posted 2022-12-20 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Sports Nutrition
Keywords: sports nutrition; survey; nutrition knowledge

STUDY DESIGN:
Intervention Model Description: Single survey, one version for student athletes survey and another version for Influencers of student athletes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Survey for student athletes (Other): 15 to 20 minute online questionnaire completed using Qualtrics
  Interventions: Other: Survey of sports nutrition knowledge
- Survey for influencers of student athletes (Other): 15 to 20 minute online questionnaire completed using Qualtrics
  Interventions: Other: Survey of sports nutrition knowledge

INTERVENTIONS:
Other: Survey of sports nutrition knowledge — Questionnaire

SUMMARY:
The objective of this testing is to gain a better understanding of sports nutrition knowledge in high school athletes and their influencers (coaches, strength and conditioning coaches, athletic therapists, dieticians). Since the sports nutrition knowledge of the high school athletes will be limited, nutrition behaviors will be assessed to infer knowledge of sports nutrition.

The secondary objective is to determine the primary sources of nutrition knowledge in these populations.

ELIGIBILITY:
Inclusion Criteria for Athletes

1. Participants are male or female between 14-19 years of age, inclusive.
2. Participants must be participating on a high school varsity team, or Amateur Athletic Union, National, or State travel team.
3. Participants must be attending high school in the United States.
4. Participant understands what is required to complete the study and signs forms providing informed consent to complete the questionnaire
5. Participant or legal guardian is able and willing to sign the Informed Consent Form.

Inclusion Criteria for Influencers

1. Participants must be currently coaching, or a practitioner for a high school varsity team, or an Amateur Athletic Union, National, or State, travel team of high school students aged (14-19 years).
2. Participants must work with/at a high school in the United States.
3. Participant understands what is required to complete the study and signs forms providing informed consent to complete the questionnaire

Exclusion Criteria for Athletes

1. Participant has a condition the Investigator believes would interfere with his or her ability to provide informed consent, which might put the individual at undue risk.
2. Participant is pregnant.

Exclusion Criteria for Influencers

1. Participant has a condition the Investigator believes would interfere with his or her ability to provide informed consent, which might put the individual at undue risk.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Better understand the level of sports nutrition knowledge of high school athletes | To complete a one-time 15 to 20 minute online questionnaire they may access at any time using a cell phone, computer, or tablet.
  Measured by determining the number of respondents that score greater than 75 percent on the sports nutrition knowledge questionnaire. A higher score is better than a lower score.
Better understand the level of sports nutrition knowledge of influencers of high school athletes | To complete a one-time 15 to 20 minute online questionnaire they may access at any time using a cell phone, computer, or tablet.
  Measured by determining the number of respondents that score greater than 75 percent on the sports nutrition knowledge questionnaire. A higher score is better than a lower score.

SECONDARY OUTCOMES:
Determine the primary sources of information for sports nutrition knowledge from high school athletes | To complete a one-time 15 to 20 minute online questionnaire they may access at any time using a cell phone, computer, or tablet.
  Measured by the sources if information selected in the survey. Credible sources of information would be better.
Determine the primary sources of information for sports nutrition knowledge from influencers of high school athletes | To complete a one-time 15 to 20 minute online questionnaire they may access at any time using a cell phone, computer, or tablet.
  Measured by the sources if information selected in the survey. Credible sources of information would be better.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Oikawa, PhD, Principal Investigator — PepsiCo, Inc. Sports Science
Locations (1):
- Remote survey, no facility visits. Survey managed by PepsiCo at IMG Academy, Bradenton, Florida, United States

IPD SHARING:
Plan to Share IPD: No